CLINICAL TRIAL: NCT06109090
Title: Influence of the Environmental Context on Neuro-psychomotor Development in Adopted Children
Acronym: ADOPT_TNPEE
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6051
Record Dates: First submitted 2023-10-13; First posted 2023-10-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Adoption
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adopted children: Patients included in the study must meet the following inclusion criteria:
  * Signing the informed consent
  * Age between 6 and 10 years
  * Adopted after the first year of life
  The exclusion criteria for this study are:
  * Comorbidity with other pathologies
  * Children adopted from birth
  * Cognitive impairment (IQ<85)
  Interventions: Other: Neuropsychological testing

INTERVENTIONS:
Other: Neuropsychological testing — In this study, the Vineland Adaptive Behavior Scale is administered, which evaluates the child's adaptive functioning, particularly in four areas: communication, socialization, daily living skills, and motor activities. The Child Behavior Checklist (CBCL) questionnaire is also administered, which is a questionnaire given to parents that highlights elements related to internalizing and externalizing behavioral disorders.
  For the assessment of executive functions, a series of tests are administered to evaluate specific functions. These tests are chosen from a list of available tests according to the document from the Italian Society of Child Neuropsychiatry, titled "Assessment of attention and executive functions in developmental age: review of Italian instruments and proposal of a battery for in-depth analysis."

SUMMARY:
The neuro-psychomotor development of children is influenced by multiple factors that play a crucial role in determining normal development or the onset of difficulties and atypicalities. Among these, the environmental context plays a fundamentally relevant role in modulating the child's abilities. Previous studies have compared children who have lived in foster care for at least 8 months with children who have always been within their own family nucleus, highlighting deficits in growth, development, and cognitive and behavioral skills in the former.

The aim of this project is to assess the effect of the environmental context on the development of executive functions and adaptive abilities in adopted children. Executive functions involve cognitive processes such as initiation, planning, organization, and regulation of behavior, while adaptive abilities include skills that allow the child to respond to demands from the external environment.

The project is conducted in two phases: a retrospective and a parallel prospective phase. The retrospective phase involves the analysis of the clinical records of adopted children in school age at the Pediatric, Child Neuropsychiatry, and Clinical Psychology units of the Fondazione Policlinico A. Gemelli IRCCS. The prospective phase consists of evaluating executive functions and adaptive abilities using specific tools recommended by the Italian Society of Child Neuropsychiatry, including the Vineland Adaptive Behavior Scales for adaptive abilities and a series of specific tests for executive functions, included in the document "Assessment of attention and executive functions in developmental age: review of Italian instruments and proposal of a battery for in-depth analysis." Additionally, to assess internalizing or externalizing behavioral aspects, parents will complete the Child Behavior Checklist (CBCL) questionnaire.

Through this study, the investigators aim to deepen the understanding of the role of the environmental context in the neuro-psychomotor development of adopted children, with particular attention to executive functions and adaptive abilities. The results obtained may provide valuable information for a better understanding of the underlying mechanisms and for the implementation of targeted interventions aimed at the optimal support of these children during their growth and development journey.

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent
* Age between 6 and 10 years
* Adopted after the first year of life

Exclusion Criteria:

* Comorbidity with other pathologies
* Children adopted from birth
* Cognitive impairment (IQ<85)

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who have had the experience of adoption in the early years of life
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
Trial making test | 10 minutes
  This test assesses various cognitive skills, including attention, visuo-motor planning, sustained attention, and working memory. Participants are given an A4 sheet with numbered circles and instructed to quickly connect them in ascending order. There are two TMT forms: TMT A with only numbers (1 to 25) and TMT B with alternating numbers and letters (1, A; 2, B; … to 13). Scarpa et al. introduced a new 'A/B' form between A and B, using only letters (A to Z), where participants connect letters in alphabetical order. This aims to ensure that children, especially younger ones, possess the alphabetical knowledge needed for part B.
  Scarpa, P et al. doi:10.1007/s10072-006-0717-5
Wisconsin Card Sorting Test | 10 minutes
  The Wisconsin Card Sorting Test (WCST) is a neuropsychological assessment of set-shifting, measuring one's ability to demonstrate flexibility in response to changes in reinforcement. Participants are presented with stimulus cards and instructed to match them. Crucially, they are not provided with explicit instructions on how to make the matches but receive feedback indicating whether their choices are correct or incorrect. In its initial release, the test involved an evaluator using paper cards, positioned on one side of the desk while the participant faced them on the other side.
Italian battery for ADHD (BIA) | 15 minutes
  Sub-test used: Stroop test/ Alternative sentence completion/ Test for the assessment of impulsive behavior
Luria's motor tasks | 15 minutes
  Motor planning and executive action control were investigated using Luria's motor tasks. In the 'contrast' task, which assessed the ability to prevent interference effects, participants were required to execute an action opposite to that performed by the examiner, resisting the inclination to imitate the examiner's action. Inhibition of control was assessed through a 'Go-No-Go' task. Scores for each subtest ranged from 0 (no correct responses) to 3 (all correct responses). The total score was the sum of the three subtest scores, with a range of 0 to 9.
  Scarpa, P et al. doi:10.1007/s10072-006-0717-5
London's tower test | 15 minutes
  The Tower of London (TOL) test, developed by Shallice in 1982 and further refined by Norman and Shallice in 1986, is one of the most widely used tools to assess strategic decision-making and problem-solving skills in children and adolescents aged 4 to 13. It serves both clinical and research purposes. The test involves a set-up with three pegs of varying lengths and three balls-red, green, and blue-that must be moved to achieve a configuration specified by the examiner. This test is instrumental in studying and measuring planning and monitoring abilities in task execution.

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scale | 10 minutes
  The Vineland assesses adaptive behavior across a wide age range, from birth to 90 years old. It comprises five main domains, each with 2-3 subdomains: Communication, Daily Living Skills, Socialization, Motor Skills, and optionally, Maladaptive Behavior. Administered individually, it features 11 general subdomains grouped into Communication, Daily Living Skills, Socialization, and Motor Skills. Subdomain scores contribute to domain composite scores, and these, in turn, combine to form adaptive behavior composites. For individuals aged 0 to 6 years 11 months, four domain composite scores are calculated, while those aged 7 to 90 have a composite based on three domains: communication, daily living skills, and socialization.
Child Behavior Checklist (CBCL) questionnaire | 10 minutes
  The Child Behavior Checklist (CBCL) is a segment of the Achenbach System of Empirically Based Assessment (ASEBA), a tool employed for identifying behavioral and emotional issues in children and adolescents. Administered by parents, the CBCL involves responding to 113 questions, with scores assigned on a three-point Likert scale (0=absent, 1=occurs sometimes, 2=occurs often).

CONTACTS AND LOCATIONS:
Overall Officials: Giorgia Coratti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy